CLINICAL TRIAL: NCT07317843
Title: Home-Based Passive Heat Therapy-Towards a Scalable Intervention to Improve Cardiovascular Health in Persons With Spinal Cord Injury
Brief Title: Home-Based Heat Therapy in Spinal Cord Injury to Improve Cardiovascular Health
Acronym: IIS_SCIDoD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002046; CDMRP-SC240010 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs (CDMRP))
Record Dates: First submitted 2025-12-18; First posted 2026-01-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: SCI - Spinal Cord Injury
Keywords: SCI; heat therapy; heat stress; passive heat; vascular function
MeSH Terms: conditions — Spinal Cord Injuries; Hyperthermia; Heat Stress Disorders | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEAT (Experimental): The experimental arm (HEAT) participants undergo an 8-week intervention with 4 weekly passive heat therapy sessions (home based for 7 of 8 weeks) using an electrical heating blanket at a temperature of 42 degrees C.
  Interventions: Other: HEAT - Passive Heat Therapy
- SHAM (Sham Comparator): For participants in SHAM, the heating blankets will be warm (~34°C) but will not reach a temperature that elevates core temperature. As in the HEAT arm, sessions will be home based for 7 of 8 weeks.
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Other: HEAT - Passive Heat Therapy — Participant rests under a heated blanket until the core body temperature has increased at minimum 1 degree Celsius. This usually takes approximately 1 hour. The intervention is performed 4 times a week for a total of 8 weeks.
  Arms: HEAT
Other: Sham (No Treatment) — The SHAM intervention participant will rest under a heated blanket that is not set to the degree that the HEAT arm receives. There is no increase of core body temperature.
  Arms: SHAM

SUMMARY:
The study is designed to investigate the effects of passive heat therapy on blood vessel health in 40 people (48 enrolled with attrition rate of 20%). Following an extensive set of vascular function tests, participants will engage in either a passive heat therapy intervention for 60 minutes, 4 times a week for 8 weeks, or a placebo intervention at a lower temperature. Seven of the 8 weeks of intervention will occur in the home setting. Vascular function tests will be repeated after the 8 weeks to determine if chronic passive heat stress improved vascular health.

DETAILED DESCRIPTION:
The experimental arm (HEAT) participants undergo an 8-week intervention with 4 weekly passive heat therapy sessions. The aim of each session is to raise the participants' core temperature by at least 1°C by resting under heating blankets set at approximately 42°C. The control arm (SHAM) participants undergo the same procedure as above except the temperature setting of the blankets is lower at approximately 34°C.

Screening, baseline assessments and the first 4 sessions will be conducted in the investigator's SCI lab to familiarize the participant with how to apply the heating blankets and ensure safety. After the 4th session, participants will receive a heating blanket for use at home in the remaining 7 intervention weeks. Cardiac MRI and peripheral vascular assessments are performed at baseline and within two weeks after completing the intervention. Weekly sessions (4x per week) in weeks 2 to 8 will be performed at home and secure VA-approved online video conferencing software will be used by study staff to remotely supervise the sessions and collect data.

ELIGIBILITY:
Inclusion Criteria:

1. Participant demonstrates understanding of the study and has provided an appropriately signed and dated informed consent.
2. Participants will be male or female, 18-60 years of age, at the time of Visit 0.
3. Female participants must be non-lactating. Female patients are eligible only if they have a negative pregnancy test throughout the study period (or are postmenopausal). Postmenopausal women taking hormone replacement will be included if they have been on a stable dose for =6 months.
4. Stable SCI (AIS A or B) of longer than 1-year duration.
5. Use of medications for clinical management of medical problems directly related to SCI is not considered an exclusion criterion. Status such as detrusor instability, muscle spasms, and other common SCI problems (other than those that could alter vascular responsiveness) may be allowed for those SCI participants who have been on stable doses for =6 months. Results from participants taking such medications will be analyzed to determine possible medication-related differences from those on no medications.

Exclusion Criteria:

1. Participants who smoke, or:
2. Uses daily administration of anti-inflammatory medications (stable doses of NSAIDs or statins are acceptable; steroids are exclusionary)
3. Uses daily administration of vasoactive medications (e.g., alpha antagonists or agonists or phosphodiesterase inhibitors).
4. Has a current pressure ulcer or skin breakdown.
5. Has an active, uncontrolled, autoimmune or inflammatory disorder
6. Has no history of or current alcohol or substance use disorder
7. Has a history of heat related illness (e.g., heat stroke)
8. Has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study. This includes, but is not limited to, a clinically relevant medical or surgical history.
9. Is unlikely to cooperate with the requirements of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Laser Doppler Flowmetry (LDF) | From baseline to end of treatment at 8 weeks
  Measure of skin blood flow due to local skin heating

SECONDARY OUTCOMES:
Endothelial Peripheral Arterial Tone (EndoPAT) | Baseline to end of treatment at 8 weeks
  Measures the changes in finger pulsatile arterial volume
Venous Occlusion Plethysmography (VOP) | From baseline to end of treatment at 8 weeks
  Limb blood flow measurement
Cardiac MRI | Baseline to end of treatment at 8 weeks
  Measures stiffness of the aorta

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Trbovich, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Audie L Murphy Veterans Memorial Hospital, South Texas Veterans Health Care System, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No